CLINICAL TRIAL: NCT02556918
Title: Sitagliptin for the Prevention and Treatment of Hyperglycemia in Patients With Type 2 Diabetes Undergoing Cardiac Surgery
Brief Title: Sitagliptin for Hyperglycemia in Patients With T2DM Undergoing Cardiac Surgery
Acronym: SITA-CABGDM
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Guillermo Umpierrez, MD, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB00082180
Record Dates: First submitted 2015-09-21; First posted 2015-09-22 (Estimated); Results first posted 2019-12-23 (Actual); Last update posted 2019-12-23 (Actual); Status verified 2019-12

CONDITIONS: Hyperglycemia
Keywords: Coronary artery bypass graft surgery (CABG); Type 2 Diabetes
MeSH Terms: conditions — Hyperglycemia; Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Insulin; Insulin Glargine; Insulin Lispro; Insulin Aspart

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sitagliptin (Experimental): Subjects undergoing cardiac surgery with type 2 diabetes (T2D) will be randomized to receive one tablet of sitagliptin once a day.Subjects with stress hyperglycemia (defined as a blood glucose (BG) greater than 180 mg/dL) in the intensive care unit (ICU) will continue to receive sitagliptin and will be started on continuous intravenous insulin (Regular Human Insulin) adjusted to achieve and maintain a BG target between 110 - 180 mg/dL following standard hospital protocol. Additionally, once moved to the regular floors and out of ICU, the subjects can receive insulin glargine, insulin lispro, and/or insulin aspart depending on the blood glucose level.
  Interventions:
  Drug: Sitagliptin Drug: Regular Human Insulin Drug: Insulin glargine Drug: Supplemental insulin (Insulin lispro) Drug: Supplemental insulin (Insulin aspart)
  Interventions: Drug: Sitagliptin; Drug: Regular Human Insulin; Drug: Insulin glargine; Drug: Supplemental insulin (Insulin lispro); Drug: Supplemental insulin (Insulin aspart)
- Placebo (Placebo Comparator): Subjects undergoing cardiac surgery with type 2 diabetes will be randomized to receive one tablet of placebo once a day.Subjects with stress hyperglycemia (defined as a blood glucose (BG) greater than 180 mg/dL) in the intensive care unit (ICU) will continue to receive a placebo and will be started on continuous intravenous insulin (Regular Human Insulin) adjusted to achieve and maintain a BG target between 110 - 180 mg/dL following standard hospital protocol. Additionally, once moved to the regular floors and out of ICU, the subjects can receive insulin glargine, insulin lispro, and/or insulin aspart depending on the blood glucose level.
  Interventions:
  Drug: Placebo Drug: Regular Human Insulin Drug: Insulin glargine Drug: Supplemental insulin (Insulin lispro) Drug: Supplemental insulin (Insulin aspart)
  Interventions: Drug: Placebo; Drug: Regular Human Insulin; Drug: Insulin glargine; Drug: Supplemental insulin (Insulin lispro); Drug: Supplemental insulin (Insulin aspart)

INTERVENTIONS:
Drug: Sitagliptin — Subjects will take one pill daily starting one day prior to surgery until discharge from the hospital. Sitagliptin will be dispensed orally at 100 mg/day for patients with a glomeruler filtration rate (GFR) greater than or equal to 50. Patients with a GFR between 30-49 will receive 50 mg/day.
  Other Names: Januvia
  Arms: Sitagliptin
Drug: Placebo — One pill daily starting one day prior to surgery until discharge from the hospital.
  Arms: Placebo
Drug: Regular Human Insulin — Continuous intravenous insulin given to intensive care unit (ICU) patients with a blood glucose (BG) greater than 180 mg/DL and will be started on Regular Human Insulin adjusted to achieve and maintain a BG target between 110 - 180 mg/dL following standard hospital protocol.Intravenous insulin infusion will be continued until the patient is able to eat and/or is transferred to non-ICU service. In previous studies, average length of insulin infusion in patients with stress hyperglycemia was 16.9±19 hours and the amount of IV insulin requirement was 18.6±24.3 U/day.
  Other Names: Novolin-R; Humulin-R
Drug: Insulin glargine — Patients that required continuous insulin infusion (CII) at a rate >1U/h will be transitioned to basal insulin (glargine/detemir). Calculate total daily dose (TDD) of insulin from the average CII rate during the last four hours of infusion (example, if the average rate is 2 U/hr., the TDD is 48 U/day) Give 50% of calculated dose as basal (glargine/detemir) insulin every day. Basal insulin will be given approx. 4 hours before discontinuation of CII.
  The total daily insulin dose will be adjusted as follow:
  Fasting and pre-meal BG between 100-180 mg/dl without hypoglycemia the previous day: no change Fasting and pre-meal BG between >180-240 mg/dl: increase basal dose by 10% every day Fasting and pre-meal BG >241 mg/dl: increase basal dose by 20% every day Fasting and pre-meal BG <100 mg/dl: stop basal
  Other Names: Lantus
Drug: Supplemental insulin (Insulin lispro) — Insulin lispro will be administered before meals in addition to scheduled insulin dose following the supplemental insulin scale protocol. At bedtime, half of supplemental sliding scale insulin starting at blood glucose (BG) greater than 240 mg/dL will be given. For the subjects receiving supplemental insulin lispro with BG levels greater than 180 mg/dL, then supplemental insulin scale is as follows:
  * BG between 181-220 mg/dL; 2-4 units of insulin lispro
  * BG between 221-260 mg/dL; 3-5 units of insulin lispro
  * BG between 261-300 mg/dL; 4-6 units of insulin lispro
  * BG between 301-350 mg/dL; 5-7 units of insulin lispro
  * BG between 351-400 mg/dL; 6-8 units of insulin lispro
  * BG greater than 400 mg/dL; 7-9 units of insulin lispro
  Other Names: Humalog
Drug: Supplemental insulin (Insulin aspart) — Insulin aspart will be administered before meals in addition to scheduled insulin dose following the supplemental insulin scale protocol. At bedtime, half of supplemental sliding scale insulin starting at blood glucose (BG) greater than 240 mg/dL will be given. For the subjects receiving supplemental insulin aspart with BG levels greater than 180 mg/dL, then supplemental insulin scale is as follows:
  * BG between 181-220 mg/dL; 2-4 units of insulin aspart
  * BG between 221-260 mg/dL; 3-5 units of insulin aspart
  * BG between 261-300 mg/dL; 4-6 units of insulin aspart
  * BG between 301-350 mg/dL; 5-7 units of insulin aspart
  * BG between 351-400 mg/dL; 6-8 units of insulin aspart
  * BG greater than 400 mg/dL; 7-9 units of insulin aspart
  Other Names: Novolog

SUMMARY:
The purpose of this study is to determine whether treatment with sitagliptin reduces the frequency and severity of high blood sugar (hyperglycemia) after cardiac surgery and to determine whether treatment with sitagliptin is effective in maintaining blood sugar control in patients with type 2 diabetes (T2D).

DETAILED DESCRIPTION:
The purpose of this study is to determine whether treatment with sitagliptin reduces the frequency and severity of high blood sugar (hyperglycemia) and the need for continuous intravenous insulin infusion (CII) in the intensive care unit (ICU) in patients with type 2 diabetes (T2D) undergoing coronary artery bypass graft (CABG) surgery. In addition, the study seeks to determine whether treatment with sitagliptin is effective in maintaining glycemic control and in preventing the need for subcutaneous (SC) insulin therapy in patients with T2D during the transition from intensive care unit (ICU) to regular floor in cardiac surgery patients with T2D.

ELIGIBILITY:
Inclusion Criteria:

* The ability to provide informed consent
* Ages 18 to 80 years old
* Male or female
* Scheduled to undergo cardiac surgery
* Type 2 Diabetes treated with diet, oral agents,

Exclusion Criteria:

* Severely impaired kidney function (glomeruler filtration rate (GFR ) less than 30 ml/min)
* Clinically significant liver failure
* Imminent risk of death (brain death or cardiac standstill)
* Gastrointestinal obstruction or adynamic ileus
* Expected to require gastrointestinal suction
* Clinically relevant pancreatic or gallbladder disease
* Using oral or injectable corticosteroid
* Mental condition rendering the subject unable to understand the nature, scope, and possible consequences of the study
* Female subjects are pregnant or breast feeding at time of enrollment into the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2016-01; Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Umpierrez, MD, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Grady Health System, Atlanta, Georgia
  - Emory Univeristy Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One participant died during hospital admission before receiving study medication.
Groups:
- Sitagliptin: Sitagliptin: Subjects will take one pill daily starting one day prior to surgery until discharge from the hospital. Sitagliptin will be dispensed orally at 100
Period: Overall Study
Arm/Group | Sitagliptin | Placebo
Started | 100 | 101
Completed | 91 | 91
Not Completed | 9 | 10
Not completed — Protocol Violation | 5 | 6
Not completed — Withdrawal by Subject | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 100 | 101 | 201
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (9.1) | 63.3 (7.8) | 63.8 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 30 | 53
  Male | 77 | 71 | 148
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 24 | 24 | 48
  White | 72 | 74 | 146
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 100 | 101 | 201

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Hyperglycemia in the Intensive Care Unit (ICU)
Description: Number of patients with blood glucose (BG) levels greater than 180 mg/dl
Time Frame: 2 days (average time of discharge from ICU)
Measure: Count of Participants; unit: Participants
Groups:
- Sitagliptin: Insulin glargine: Patients that required continuous insulin infusion (CII) at a rate >1U/h will be transitioned to basal insulin (glargine/detemir). Calculate total daily dose (TDD) of insulin from the average CII rate during the last four hours of infusion (example, if the average rate is 2 U/hr., the TDD is 48 U/day)
  Supplemental insulin (Insulin aspart): Insulin aspart will be administered before meals in addition to scheduled insulin dose following the supplemental insulin scale protocol.
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
Participants | 76 | 68

2. Primary Outcome: Number of Patients With Persistent Hyperglycemia
Description: Number of patients with two consecutive fasting and/or pre-meal blood glucose (BG) greater than 180 mg/dl, or with average daily BG greater than 80 mg/dl who require rescue therapy with subcutaneous (SC) insulin after discontinuation of continuous intravenous insulin infusion (CII).
Time Frame: 10 days (average time of discharge from the hospital)
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
Participants | 58 | 59

3. Secondary Outcome: Number of Patients Requiring Continuous Intravenous Insulin Infusion (CII)
Description: Number of patients requiring CII to achieve a blood glucose level (BG) target between 150-200 mg/dl
Time Frame: 2 days (average time of discharge from ICU)
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
Participants | 86 | 85

4. Secondary Outcome: Mean Blood Glucose (BG) Concentration in the Intensive Care Unit (ICU)
Description: Mean blood glucose (BG) concentration of ICU patients during recovery period.
Time Frame: 2 days (average time of discharge from ICU)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
mmol/L | 148.7 (15.8) | 149.8 (16.0)

5. Secondary Outcome: Total IV Insulin in ICU
Description: Total IV insulin in ICU during recovery period.
Time Frame: 2 days (average time of discharge from ICU)
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
units | 100.43 (123.44) | 95.68 (118.32)

6. Secondary Outcome: Mean Insulin Dose Per Day During Intensive Care Unit (ICU) Recovery
Description: Mean insulin infusion dose per day of ICU patients during recovery period.
Time Frame: 2 days (average time of discharge from ICU)
Measure: Mean (Standard Deviation); unit: unit/day
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
unit/day | 45.9 (36.1) | 46.4 (36.0)

7. Secondary Outcome: Duration of Continuous Intravenous Insulin Infusion (CII)
Description: Total hours of continuous intravenous insulin infusion (CII)
Time Frame: Up to 48 hours (average time of discharge from ICU)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
hours | 27.7 (27.6) | 27.7 (28.0)

8. Secondary Outcome: Number of Patients Requiring Subcutaneous (SQ) Insulin After Discontinuation of Continuous Intravenous Insulin Infusion (CII)
Description: Number of patients requiring subcutaneous (SQ) insulin after discontinuation of continuous intravenous insulin infusion (CII)
Time Frame: 10 days (average time of discharge from the hospital)
Population: Some patients were not transitioned to SQ insulin because they stayed on CII due to complications, these patients were taken off the analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 87 | 86
Participants | 74 | 78

9. Secondary Outcome: Median Number of Days of Subcutaneous (SC) Insulin After Discontinuation of Continuous Intravenous Insulin Infusion (CII)
Description: Median number of days patients requiring SC insulin after discontinuation of CII
Time Frame: Up to 14 days (time of discharge from the hospital)
Population: as for outcome 8
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 87 | 86
days | 4 [0 to 14] | 4 [0 to 10]

10. Secondary Outcome: Mean Post-operative Blood Glucose (BG) Concentration
Description: Mean post-operative blood glucose (BG) concentration during recovery period.
Time Frame: 10 days (average time of discharge from the hospital)
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
mmol/L | 154.2 (29.0) | 156.5 (36.1)

11. Secondary Outcome: Amount of Subcutaneous (SC) Insulin Taken in Intensive Care Unit (ICU)
Description: Total amount of SC insulin taken by ICU patients during recovery period.
Time Frame: 2 days (average time of discharge from ICU)
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
units | 1.0 (6.4) | 2.2 (13.1)

12. Secondary Outcome: Amount of Subcutaneous (SC) Insulin in Intensive Care Unit (ICU) 48 Hours
Description: Amount of subcutaneous (SC) insulin in intensive care unit (ICU) 48 hours during recovery period.
Time Frame: 48 hours during recovery period
Measure: Mean (Standard Deviation); unit: units
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
units | 0.48 (3.8) | 1.5 (8.7)

13. Secondary Outcome: Number of Subjects With Hyperglycemia in Intensive Care Unit (ICU)
Description: Number of subjects with hyperglycemia (blood glucose greater than or equal to 300 mg/dL) in ICU recovery period.
Time Frame: 2 days (average time of discharge from ICU)
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
Participants | 5 | 3

14. Secondary Outcome: Number of Subjects With Hyperglycemia (Blood Glucose Greater Than or Equal to 300 mg/dL) in Non-ICU
Description: Number of subjects with hyperglycemia (blood glucose greater than or equal to 300 mg/dL) in non-ICU recovery period.
Time Frame: 10 days (average time of discharge from the hospital)
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
Participants | 20 | 12

15. Secondary Outcome: Number of Patients With Hypoglycemic Events in Intensive Care Unit (ICU)
Description: Number of patients with events (blood glucose less than 70 mg/dL) in patients in intensive care unit (ICU).
Time Frame: 2 days (average time of discharge from ICU)
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
Participants | 8 | 6

16. Secondary Outcome: Number of Patients With Hypoglycemic Events in Non-intensive Care Unit (ICU)
Description: Number of Patients With hypoglycemic events (blood glucose less than 70 mg/dL) in patients in non-intensive care unit (ICU).
Time Frame: 10 days (average time of discharge from the hospital)
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
Participants | 8 | 8

17. Secondary Outcome: Number of Patients With Severe Hypoglycemic Events in Intensive Care Unit (ICU)
Description: Number of Patients With severe hypoglycemia (blood glucose less than 40 mg/dL) in patients in intensive care unit (ICU).
Time Frame: 2 days (average time of discharge from ICU)
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
Participants | 0 | 0

18. Secondary Outcome: Number of Patients With Severe Hypoglycemic Events in Non-intensive Care Unit (ICU)
Description: Number of Patients With hypoglycemic events (blood glucose less than 40 mg/dL) in patients in non-intensive care unit (ICU).
Time Frame: 10 days (average time of discharge from the hospital)
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
Participants | 0 | 0

19. Secondary Outcome: Composite of Perioperative Complications
Description: Number of perioperative complications including hospital mortality, infection,acute renal failure, and acute mycordial infarction.
Time Frame: 10 days (average time of discharge from the hospital)
Measure: Number; unit: events
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
events | 63 | 42

20. Secondary Outcome: Duration of Intubation
Description: Duration that patients required to be intubated
Time Frame: 10 days (average time of discharge from the hospital)
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
days | 0.5 (1.1) | 0.7 (1.9)

21. Secondary Outcome: Length of Intensive Care Unit (ICU) Stay
Description: Total number of days spent in intensive care unit (ICU)
Time Frame: 2 days (average time of discharge from ICU)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
days | 2.0 [1.0 to 3.2] | 2.2 [1.4 to 3.9]

22. Secondary Outcome: Total Length of Hospital Stay
Description: Total number of days spent in hospital
Time Frame: 10 days (average time of discharge from the hospital)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
days | 9 [6 to 12] | 7 [6 to 13]

23. Secondary Outcome: Number of Intensive Care Unit (ICU) Readmission
Description: Number of re-admissions to intensive care unit during the same hospital course.
Time Frame: 10 days (average time of discharge from the hospital)
Measure: Number; unit: readmissions
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
readmissions | 14 | 7

24. Secondary Outcome: Number of Cerebrovascular Events
Description: Number of cerebrovascular events including permanent stroke and reversible ischemic neurologic deficit
Time Frame: 10 days (average time of discharge from the hospital)
Measure: Number; unit: events
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
events | 5 | 7

25. Secondary Outcome: Number of Subjects Readmitted to the Hospital
Description: Number of subjects readmitted to the hospital within 30 days (all-cause).
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
Participants | 10 | 12

26. Secondary Outcome: Number of Subjects Returning to the ER Within 30 Days
Description: Number of subjects returning to the ER within 30 days (all-cause).
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 91 | 91
Participants | 61 | 57

ADVERSE EVENTS:
Time Frame: one month
Arm/Group | Sitagliptin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/100 | 1/101
Serious Adverse Events (participants affected / at risk) | 80/100 | 69/101
Other Adverse Events (participants affected / at risk) | 6/100 | 5/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=100) | Placebo (N=101)
Miocardial Infarction (Cardiac disorders) | 3 (3) | 2 (3)
Cardiogenic shock (Cardiac disorders) | 1 (1) | 0 (0)
Atrial Fibrillation (Cardiac disorders) | 27 (66) | 25 (50)
Ventricular Fibrillation (Cardiac disorders) | 2 (3) | 4 (5)
Stroke (Vascular disorders) | 5 (5) | 2 (7)
Acute Kidney Injury (Renal and urinary disorders) | 20 (57) | 16 (34)
Re-admittion to ICU (General disorders) | 7 (14) | 5 (7)
Re-intubation (General disorders) | 4 (6) | 2 (2)
Surgical Site Bleeding (Vascular disorders) | 1 (1) | 1 (1)
Readmission due to surgical site infection (Infections and infestations) | 3 (3) | 5 (5)
Hospital readmissions for other reasons (General disorders) | 7 (7) | 7 (7)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=100) | Placebo (N=101)
Headache (General disorders) | 1 (1) | 1 (1)
Loss of appetite (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-05): https://cdn.clinicaltrials.gov/large-docs/18/NCT02556918/Prot_SAP_000.pdf